CLINICAL TRIAL: NCT02509156
Title: A Phase I, First-in-Human, Multicenter, Randomized, Double-Blinded, Placebo-Controlled Study of the Safety and Efficacy of Allogeneic Mesenchymal Stem Cells in Cancer Survivors With Anthracycline-Induced Cardiomyopathy
Brief Title: Stem Cell Injection in Cancer Survivors
Acronym: SENECA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Barry R Davis, Professor of Biostatistics, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-SPH-15-0443; 5UM1HL087318 (NIH)
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Cardiomyopathy Due to Anthracyclines
Keywords: Cardiomyopathy; AIC; Anthracyclines; Chemotherapy; Allogeneic; Mesenchymal stem cells; MSCs; Cancer survivors; Breast Cancer; Leukemia; Lymphoma; Sarcoma
MeSH Terms: conditions — Cardiomyopathies; Breast Neoplasms; Leukemia; Lymphoma; Sarcoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allo-MSCs (Experimental): Target dose of 100 million allo-MSCs
  Interventions: Biological: Allo-MSCs
- Placebo (Placebo Comparator): Buminate solution
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Allo-MSCs — 20 transendocardial injections of 0.4ml allo-MSCs administered to the left ventricle via NOGA Myostar injection catheter (single procedure)
  Other Names: Allogeneic Mesenchymal Stem Cells
  Arms: Allo-MSCs
Biological: Placebo — 20 transendocardial injections of 0.4ml Buminate solution administered to the left ventricle via NOGA Myostar injection catheter (single procedure)
  Other Names: Buminate solution
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to examine the safety and feasibility of delivering allogeneic human mesenchymal stem cells (allo-MSCs) by transendocardial injection to cancer survivors with left ventricular (LV) dysfunction secondary to anthracycline-induced cardiomyopathy (AIC).

The secondary purpose of this study is to obtain preliminary evidence for therapeutic efficacy of allo-MSCs delivered by transendocardial injection to cancer survivors with LV dysfunction secondary to AIC.

DETAILED DESCRIPTION:
This phase I, randomized, placebo-controlled, trial will evaluate the safety and feasibility of allo-MSCs administered by transendocardial injection in thirty-seven subjects with anthracycline-induced cardiomyopathy (AIC). The first six subjects received allo-MSC therapy (open label) and were assessed for safety and feasibility of the study procedures. Following 1 month data review of each of the six subjects by the National Heart, Lung, and Blood Institute Gene and Cell Therapy Data Safety Monitoring Board; this was followed by a randomized, double-blind clinical trial enrolling thirty-one subjects. These subjects were randomized 1:1 to receive allo-MSCs or placebo. All subjects underwent cardiac catheterization and study product administration using the NOGA Myostar catheter injection system. Subjects are being followed at 1 day, 1 week, 1 month, 6 months, and 12 months post study product injection. All endpoints are assessed at the 6 and 12 month visits which will occur 180 ±30 days and 365 ±30 days, respectively, after the day of study product injection (Day 0). For the purpose of the safety evaluations and endpoint analysis, the Investigators will utilize an "intention-to-treat" study population. In addition, because this phase I study is the first cell therapy study in this population, at 12 months available standard-of-care medical records for cancer surveillance will be reviewed for cancer recurrence.

ELIGIBILITY:
Inclusion Criteria

To participate, a subject MUST:

1. Be ≥ 18 and < 80 years of age
2. Be a cancer survivor with diagnosis of AIC
3. Have an LVEF ≤ 45% by cMRI
4. Be in NYHA class II-III
5. Have received the initial diagnosis of AIC at least six months earlier and be on stable, optimally-tolerated therapy with beta-blockers, ACE inhibitors/ARBs, and/or aldosterone antagonists for 3 months, unless contraindicated
6. Have a period of at least two years of clinical cancer-free state* and low likelihood of recurrence (a five-year risk of recurrence estimated at 30% or less), as determined by an oncologist, based on tumor type, response to therapy, and negative metastatic work-up at the time of diagnosis (*exceptions to this are carcinoma in situ or fully resected basal and squamous cell cancer of the skin.)
7. Be a candidate for cardiac catheterization

Exclusion Criteria

To participate, a subject MUST NOT HAVE:

1. A life expectancy <12 months
2. A CT scan or baseline cardiac MRI showing new tumor or suspicious lymphadenopathy raising concern of malignancy
3. Presence of obstructive CAD as determined via imaging within 5 years prior to study enrollment provided there have been no symptoms or evidence of CAD since the test
4. Had a previous myocardial infarction
5. A history of radiation therapy AND evidence of constrictive physiology and/or evidence of other patterns of non-ischemic cardiomyopathy on cardiac MRI (e.g., amyloidosis, sarcoidosis, hemochromatosis, pure radiation-induced cardiomyopathy, etc.) not consistent with AIC being the dominant etiology of heart failure
6. Valvular heart disease including 1) mechanical or bioprosthetic heart valve; or 2) severe valvular (any valve) insufficiency/regurgitation within 12 months of consent.
7. Aortic stenosis with valve area ≤ 1.5cm2
8. A history of LV reduction surgery or cardiomyoplasty
9. Evidence of cardiogenic shock
10. A history of ischemic or hemorrhagic stroke within 90 days of baseline testing
11. Liver dysfunction during baseline testing, as evidenced by enzymes (e.g., AST, ALT, alkaline phosphatase) greater than 3 times upper limit of normal
12. Diabetes with poorly controlled blood glucose levels (HbA1c > 8.5%)
13. An underlying autoimmune disorder or current immunosuppressive therapy (e.g., chronic corticosteroid, rheumatologic or immune modulating therapy) or likelihood of use of immunosuppressive therapy during participation in the trial (medications will be considered on a case by case basis)
14. A baseline eGFR <35 ml/min/1.73m2
15. A contrast allergy that cannot adequately be managed by premedication
16. Received gene or cell-based therapy from any source within the previous 12 months
17. A hematologic abnormality during baseline testing as evidenced by hemoglobin < 9 g/dl; hematocrit < 30%; absolute neutrophil count < 2,000 or total WBC count more than 2 times upper limit of normal; or platelet values < 100,000/ul
18. Evidence of active systemic infection at time of study product delivery
19. HIV and/or active HBV or HCV
20. Coagulopathy (INR > 1.5) not due to a reversible cause (e.g., warfarin and/or Factor Xa inhibitors) (see Section 6.4 re: injection procedure and anticoagulation therapy) Note: Subjects who cannot be withdrawn from anticoagulation will be excluded.
21. Presence of LV thrombus
22. Presence of a pacemaker and/or ICD generator with any of the following limitations/conditions:

    * manufactured before the year 2000
    * leads implanted < 6 weeks prior to consent
    * non-transvenous epicardial or abandoned leads
    * subcutaneous ICDs
    * leadless pacemakers
    * any other condition that, in the judgment of device-trained staff, would deem an MRI contraindicated
23. Pacemaker-dependence with an ICD (Note: pacemaker-dependent candidates without an ICD are not excluded)
24. A cardiac resynchronization therapy (CRT) device implanted < 3 months prior to consent
25. Other MRI contraindications (e.g. patient body habitus incompatible with MRI)
26. An appropriate ICD firing or anti-tachycardia pacing (ATP) for ventricular fibrillation or ventricular tachycardia within 30 days of consent
27. Ventricular tachycardia ≥ 20 consecutive beats without an ICD within 3 months of consent, or symptomatic Mobitz II or higher degree atrioventricular block without a functioning pacemaker within 3 months of consent
28. A history of drug abuse (use of illegal "street" drugs except marijuana, or prescription medications not being used appropriately for a pre-existing medical condition) or alcohol abuse (≥ 5 drinks/day for ˃ 3 months), or documented medical, occupational, or legal problems arising from the use of alcohol or drugs within the past 24 months
29. Cognitive or language barriers that prohibit obtaining informed consent or any study elements (interpreter permitted)
30. Participation (currently or within the previous 30 days) in a cardiac related investigational therapeutic (including stem cell based therapies) or device trial
31. Pregnancy, lactation, plans to become pregnant in the next 12 months, or is unwilling to use acceptable forms of birth control during study participation
32. Any other condition that, in the judgment of the Investigator or Sponsor, would be a contraindication to enrollment, study product administration, or follow-up

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Simari, MD, Study Chair — CCTRN Steering Committee Chair
Locations (7):
- United States (7):
  - Stanford University School of Medicine, Stanford, California
  - University of Florida-Department of Medicine, Gainesville, Florida
  - University of Miami-Interdiciplinary Stem Cell Institute, Miami, Florida
  - Indiana Center for Vascular Biology and Medicine, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Texas Heart Institute, Houston, Texas

REFERENCES:
- [Background] Psaltis PJ, Carbone A, Nelson AJ, Lau DH, Jantzen T, Manavis J, Williams K, Itescu S, Sanders P, Gronthos S, Zannettino AC, Worthley SG. Reparative effects of allogeneic mesenchymal precursor cells delivered transendocardially in experimental nonischemic cardiomyopathy. JACC Cardiovasc Interv. 2010 Sep;3(9):974-83. doi: 10.1016/j.jcin.2010.05.016. PMID 20850099
- [Background] Nazarian S, Halperin HR. How to perform magnetic resonance imaging on patients with implantable cardiac arrhythmia devices. Heart Rhythm. 2009 Jan;6(1):138-43. doi: 10.1016/j.hrthm.2008.10.021. Epub 2008 Oct 22. No abstract available. PMID 19121814
- [Background] Bolli R, Hare JM, Henry TD, Lenneman CG, March KL, Miller K, Pepine CJ, Perin EC, Traverse JH, Willerson JT, Yang PC, Gee AP, Lima JA, Moye L, Vojvodic RW, Sayre SL, Bettencourt J, Cohen M, Ebert RF, Simari RD; Cardiovascular Cell Therapy Research Network (CCTRN). Rationale and Design of the SENECA (StEm cell iNjECtion in cAncer survivors) Trial. Am Heart J. 2018 Jul;201:54-62. doi: 10.1016/j.ahj.2018.02.009. Epub 2018 Apr 4. PMID 29910056
- See also: Cardiovascular Cell Therapy Research Network — http://www.cctrn.org
- See also: National Heart, Lung, and Blood Institute — http://www.nhlbi.nih.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place at seven CCTRN centers between September 2016 and October 2018. The main centers are located in Texas, Florida (2 locations), Minnesota, Kentucky, Indiana, and California. Recruitment methods included www.clinicaltrials.gov, cancer survivorship organization websites, and local cancer center physician outreach.
Pre-assignment Details: 46 subjects consented to participate; 37 completed baseline testing and met eligibility criteria. This includes 6 (open label) and 31 (randomized) subjects. Reasons for failed eligibility (n=9) include elevated LVEF, failure to complete baseline testing, MRI contraindications, and investigator discretion.
Period: Open-Label Lead-In Phase
Arm/Group | Allo-MSCs | Placebo
Started | 6 | 0
Completed | 6 | 0
Not Completed | 0 | 0
Period: Randomized Phase
Arm/Group | Allo-MSCs | Placebo
Started | 14 (Includes randomized participants only) | 17
Completed | 12 | 16
Not Completed | 2 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allo-MSCs | Placebo | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (12.8) | 58.2 (11.2) | 56.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 12 | 13 | 25
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 8 | 13 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 14 | 17 | 31
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (9) | 30.4 (6.5) | 30.3 (7.6)
Heart rate [Mean (Standard Deviation); unit: beats per minute] | 74.4 (9) | 76.1 (11.2) | 75.4 (10.1)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 118.6 (21.6) | 115.4 (11.0) | 116.8 (16.4)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 68.9 (18.6) | 67.1 (11.2) | 67.9 (14.7)
Diabetes [Count of Participants; unit: Participants] | 3 | 5 | 8
Hypertension [Count of Participants; unit: Participants] | 6 | 10 | 16
Smoking (lifetime) [Count of Participants; unit: Participants] | 5 | 3 | 8
Left ventricular ejection fraction [Mean (Standard Deviation); unit: percentage of blood ejected] | 33.7 (3.4) | 32.5 (6.5) | 33.0 (5.3)
Previous hospitalization for heart failure [Count of Participants; unit: Participants] | 7 | 8 | 15
Previous emergency department visit for heart failure [Count of Participants; unit: Participants] | 4 | 3 | 7
Time since AIC diagnosis [Mean (Standard Deviation); unit: years] — Time since anthracycline induced cardiomyopathy diagnosis (years)
  years | 6.1 (5.9) | 8.7 (5.0) | 7.5 (5.5)
New York Heart Association class II [Count of Participants; unit: Participants] — Physicians use the NYHA classification system to place patients in one of four categories based on how much they are limited during physical activity. Class II is characterized by slight limitation of physical activity. The patient is comfortable at rest, however ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Participants | 13 | 13 | 26
New York Heart Association class III [Count of Participants; unit: Participants] — Physicians use the NYHA classification system to place patients in one of four categories based on how much they are limited during physical activity. Class III is characterized by marked limitation of physical activity. The patient is comfortable at rest. Less than ordinary activity however, causes fatigue, palpitation, or dyspnea.
  Participants | 1 | 4 | 5
Presence of a cardiac device [Count of Participants; unit: Participants] — Presence of a cardiac device (implantable cardioverter defibrillator or pacemaker)
  Participants | 6 | 12 | 18
Angina [Count of Participants; unit: Participants] | 3 | 5 | 8
Sustained ventricular arrhythmia [Count of Participants; unit: Participants] | 5 | 7 | 12
Leukemia [Count of Participants; unit: Participants] | 3 | 0 | 3
Breast cancer [Count of Participants; unit: Participants] | 6 | 9 | 15
Hodgkin's disease [Count of Participants; unit: Participants] | 0 | 1 | 1
Non-Hodgkin's lymphoma [Count of Participants; unit: Participants] | 1 | 5 | 6
Sarcomas [Count of Participants; unit: Participants] | 1 | 0 | 1
Multiple cancers [Count of Participants; unit: Participants] | 3 | 2 | 5
Doxorubicin [Count of Participants; unit: Participants] | 11 | 17 | 28
Epirubicin [Count of Participants; unit: Participants] | 1 | 0 | 1
Daunorubicin [Count of Participants; unit: Participants] | 2 | 0 | 2
AIC exposure [Mean (Standard Deviation); unit: mg/m^2] — Population: Limited information due to treatment record availability (>15yrs). Dosing information (mg/m^2) not always available. Data represents a subset of the cohort.
  mg/m^2
    number analyzed (Participants) | 10 | 10 | 20
    (all) | 353.0 (351.3) | 339.5 (113.6) | 346.2 (254.2)
Time from Cancer Diagnosis [Mean (Standard Deviation); unit: years] — Time from earliest diagnosis requiring anthracycline treatment
  years | 16.4 (9.5) | 18.8 (8.5) | 17.7 (8.9)
Time from last anthracycline treatment [Mean (Standard Deviation); unit: years] | 13.3 (9.3) | 16.8 (7.6) | 15.2 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Major Adverse Cardiac Events (MACE)
Description: Proportion of adjudicated events including death, hospitalization for worsening heart failure, and/or other exacerbation of heart failure (non-hospitalization).
Time Frame: Baseline to 12 months
Population: Population for safety and feasibility measures include open label lead-in participants (n=6) as well as randomized subjects (n=31).
Measure: Number; unit: events
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 20 | 17
events | 3 | 6

2. Primary Outcome: Proportion of Other Significant Clinical Events
Description: Proportion of other significant adjudicated clinical events including: non-fatal stroke, non-fatal MI, coronary artery revascularization, ventricular tachycardia/fibrillation, pericardial tamponade, infectious myocarditis, hypersensitivity reaction, neoplasm, and/or other potential deleterious late effects.
Time Frame: Baseline to 12 months
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 20 | 17
events | 0 | 1

3. Primary Outcome: Subjects With Events Precluding Their Receipt of Product
Description: Number and percent of subjects with events between randomization and study product injection (SPI) that preclude the subject from receiving product.
Time Frame: Randomization to SPI
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 20 | 17
Participants | 0 | 1

4. Primary Outcome: Subjects Who Receive Less Than 20 Injections During SPI
Description: Number and percent of subjects who receive less than 20 injections during SPI
Time Frame: During SPI procedure
Population: Population for safety and feasibility measures include open label lead-in participants (n=6) as well as randomized subjects who were participating at the time of study product injection (n=30). Note: one placebo patient withdrew after randomization but prior to injection visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 20 | 16
Participants | 1 | 0

5. Primary Outcome: Subjects Who Did Not Receive the Study Product (Either 100 Million Cells or Placebo)
Description: Number and percent of subjects who did not receive the study product (either 100 million cells or placebo)
Time Frame: During SPI procedure
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 20 | 16
Participants | 0 | 0

6. Primary Outcome: Subjects Who Have at Least One Cardiac MRI Endpoint Measure That is Uninterpretable
Description: Number and percent of subjects who have at least one cardiac MRI endpoint measure that is uninterpretable due to issues related to the device, including, but not limited to, inability to undergo the procedure.
Time Frame: Baseline to 12 months
Population: Population for safety and feasibility measures include open label lead-in participants (n=6) as well as randomized subjects (n=31). Analysis population includes only participants who completed an MRI at 12 months (n=32).
Measure: Count of Participants; unit: Participants
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 18 | 14
Participants | 1 | 4

7. Primary Outcome: Subjects Who Fail to Complete Follow-up
Description: Number and percent of subjects who fail to complete follow up
Time Frame: Baseline to 12 months
Population: Population for safety and feasibility analysis include open label lead-in participants (n=6)
Measure: Count of Participants; unit: Participants
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 20 | 17
Participants | 2 | 1

8. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF)
Description: Change in left ventricular ejection fraction as assessed via cardiac MRI.
Time Frame: Baseline to 12 months
Population: Participants who had available analyzable LVEF at baseline and 12 month.
Measure: Mean (Standard Deviation); unit: percentage of end diastolic volume
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 13
percentage of end diastolic volume | 3.47 (6.00) | 2.68 (6.85)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; Test type: Superiority; p = 0.746, ANCOVA; The change in LVEF was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.80, 95% CI 2-sided [-4.52 to 6.11], Standard Error of Mean 2.57 — Confidence intervals based on t-test

9. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF)-Trajectory
Description: The change in this measure over time is assessed using a repeated measures linear regression model of trajectory (change over time). If there is no interaction between change over time and treatment a single calculated value is the slope (the change per six months) from the model. If there is an interaction, the p-value for interaction is presented along with two calculated values representing the slope (the change per six months) for each treatment arm from the model.
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had available analyzable LVEF at baseline, 6 month, and 12 month.
Measure: Least Squares Mean (Standard Error); unit: percentage of end diastolic volume
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 13
percentage of end diastolic volume | 1.81 (0.86) | 1.33 (0.95)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; Repeated-measures linear regression models were used to address trajectories (upward or downward trends) over time within each of the treatment groups. If there was no significant interaction, only one trajectory (slope) was reported; Test type: Superiority; p = 0.024, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase I trial; slope of time = 1.53, Standard Error of Mean 0.63 — "Standard error of the mean" is the standard error of the estimate of the slope of time

10. Secondary Outcome: Change From Baseline in Global Strain (HARP MRI)
Description: Change in global circumferential strain as assessed via cardiac MRI
Time Frame: Baseline to 12 months
Population: Participants with available analyzable global circumferential strain at baseline and 12 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 11 | 13
percent | -0.83 (1.70) | -0.12 (2.86)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; The change in global strain was compared using ANCOVA analyses adjusting for baseline values; Test type: Superiority; p = 0.328, ANCOVA; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-2.68 to 1.26], Standard Error of Mean 0.94 — Confidence intervals based on t-test

11. Secondary Outcome: Change From Baseline in Global Strain (HARP MRI)-Trajectory
Description: as for outcome 9
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had available analyzable global strain at baseline, 6 month, and 12 month.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 11 | 13
percent | -0.49 (0.24) | -0.04 (0.36)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.261, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase I trial; slope of time = -0.26, Standard Error of Mean 0.23 — "Standard error of the mean" is the standard error of the estimate over time of the slope

12. Secondary Outcome: Change From Baseline in Regional Strain (HARP MRI)
Description: Change in regional longitudinal strain as assessed via cardiac MRI
Time Frame: Baseline to 12 months
Population: Participants with available analyzable regional longitudinal strain at baseline and 12 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 13
percent | -1.20 (3.34) | 0.38 (3.73)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; The change in regional strain was compared using ANCOVA analyses adjusting for baseline values; Test type: Superiority; p = 0.071, ANCOVA; Mean Difference (Final Values) = -1.58, 95% CI 2-sided [-4.51 to 1.35], Standard Error of Mean 1.41 — Confidence intervals based on t-test

13. Secondary Outcome: Change From Baseline in Regional Strain (HARP MRI)-Trajectory
Description: as for outcome 9
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had available analyzable regional strain at baseline, 6 month, and 12 month.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 13
percent | -0.58 (0.42) | 0.21 (0.52)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.689, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase I trial; slope of time = -0.14, Standard Error of Mean 0.35 — "Standard error of the mean" is the standard error of the estimate over time of the slope

14. Secondary Outcome: Change From Baseline in Left Ventricular End Diastolic Volume Index (LVEDVI)
Description: Change in left ventricular end diastolic volume index as measured via cardiac MRI
Time Frame: Baseline to 12 months
Population: Participants with available analyzable LVEDVI at baseline and 12 months
Measure: Mean (Standard Deviation); unit: ratio- unitless
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 13
ratio- unitless | -2.30 (16.97) | -3.36 (15.18)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; The change in LVEDVI was compared using ANCOVA analyses adjusting for baseline values; Test type: Superiority; p = 0.935, ANCOVA; Mean Difference (Final Values) = 1.06, 95% CI 2-sided [-12.33 to 14.45], Standard Error of Mean 6.46 — Confidence intervals based on t-test

15. Secondary Outcome: Change From Baseline in Left Ventricular End Diastolic Volume Index (LVEDVI)-Trajectory
Description: as for outcome 9
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had available analyzable LVEDVI at baseline, 6 month, and 12 month.
Measure: Least Squares Mean (Standard Error); unit: ratio-unitless
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 13
ratio-unitless | -0.94 (2.38) | -1.98 (1.95)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.325, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase I trial; slope of time = -1.56, Standard Error of Mean 1.55 — "Standard error of the mean" is the standard error of the estimate over time of the slope

16. Secondary Outcome: Change From Baseline in Left Ventricular End Systolic Volume Index (LVESVI)
Description: Change in left ventricular end systolic volume index as assessed via cardiac MRI
Time Frame: Baseline to 12 months
Population: Participants with available analyzable LVESVI at baseline and 12 months
Measure: Mean (Standard Deviation); unit: ratio- unitless
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 13
ratio- unitless | -3.62 (15.66) | -4.28 (14.18)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; The change in LVESVI was compared using ANCOVA analyses adjusting for baseline values; Test type: Superiority; p = 0.919, ANCOVA; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-11.75 to 13.08], Standard Error of Mean 5.99 — Confidence intervals based on t-test

17. Secondary Outcome: Change From Baseline in Left Ventricular End Systolic Volume Index (LVESVI)-Trajectory
Description: as for outcome 9
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had available analyzable LVESVI at baseline, 6 month, and 12 month.
Measure: Least Squares Mean (Standard Error); unit: ratio- unitless
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 13
ratio- unitless | -2.05 (2.14) | -2.34 (1.81)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.183, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase I trial; slope of time = -1.99, Standard Error of Mean 1.45 — "Standard error of the mean" is the standard error of the estimate over time of the slope

18. Secondary Outcome: Change From Baseline in Left Ventricular Sphericity Index
Description: Change in Left Ventricular Sphericity Index as assessed by cardiac MRI. Sphericity index is the ratio of the long and short axis measurements of the left ventricle.
Time Frame: Baseline to 12 months
Population: Participants who had available analyzable LV sphericity index at baseline and 12 month LV.
Measure: Mean (Standard Deviation); unit: ratio- unitless
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 13
ratio- unitless | 0.01 (0.08) | -0.07 (0.09)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; The change in LV sphericity index was compared using ANCOVA analyses adjusting for baseline values; Test type: Superiority; p = 0.124, ANCOVA; Mean Difference (Final Values) = 0.077, 95% CI 2-sided [0.003 to 0.15], Standard Error of Mean 0.035 — Confidence intervals based on t-test

19. Secondary Outcome: Change From Baseline in Left Ventricular Sphericity Index-Trajectory
Description: The change in this measure over time is assessed using a repeated measures linear regression model of trajectory (change over time). If there is no interaction between change over time and treatment a single calculated value is the slope (the change per six months) from the model. If there is an interaction, the p-value for interaction is presented along with two calculated values representing the slope (the change per six months) for each treatment arm from the model.
  Sphericity index is the ratio of the long and short axis measurements of the left ventricle.
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had available analyzable sphericity index at baseline, 6 month, and 12 month.
Measure: Least Squares Mean (Standard Error); unit: ratio-unitless
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 13
ratio-unitless | 0.005 (0.013) | -0.037 (0.012)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; Repeated-measures linear regression models were used to address trajectories (upward or downward trends) over time within each of the treatment groups. A time by treatment interaction was assessed; Test type: Superiority; There was a significant treatment and time interaction (p=0.024), so we report a slope for each treatment arm

20. Secondary Outcome: Change From Baseline in Area of Injury
Description: Change in the scar percent (scar mass normalized to left ventricular mass) as assessed via cardiac MRI.
Time Frame: Baseline to 12 months
Population: Participants who had available analyzable scar percent at baseline and 12 month.
Measure: Mean (Standard Deviation); unit: percentage of mass
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 11 | 10
percentage of mass | -1.06 (2.44) | -0.41 (2.76)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; The change in scar percent was compared using ANCOVA analyses adjusting for baseline values; Test type: Superiority; p = 0.993, ANCOVA; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-3.05 to 1.74], Standard Error of Mean 1.14 — Confidence intervals based on t-test

21. Secondary Outcome: Change From Baseline in Area of Injury-Trajectory
Description: as for outcome 9
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had available analyzable scar percent at baseline, 6 month, and 12 month.
Measure: Least Squares Mean (Standard Error); unit: percentage of mass
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 11 | 10
percentage of mass | -0.56 (0.41) | -0.27 (0.43)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.151, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase I trial; slope of time = -0.44, Standard Error of Mean 0.29 — "Standard error of the mean" is the standard error of the estimate over time of the slope

22. Secondary Outcome: Change From Baseline in Exercise Tolerance (Six Minute Walk Test)
Description: Change in the distance walked (in meters) as measured by the six minute walk test. Two walk tests were completed at each endpoint visit (separated by 30 min). The average distance of the two walk tests will be used for analysis.
Time Frame: Baseline to 12 months
Population: Participants who had available analyzable walk tests at baseline and 12 month.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 15
meters | 34.96 (61.62) | -3.07 (42.90)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; The change in distance walked was compared using ANCOVA analyses adjusting for baseline values; Test type: Superiority; p = 0.056, ANCOVA; Mean Difference (Final Values) = 38.03, 95% CI 2-sided [-5.84 to 81.89], Standard Error of Mean 20.96 — Confidence intervals based on t-test

23. Secondary Outcome: Change From Baseline in Exercise Tolerance (Six Minute Walk Test)-Trajectory
Description: Change in the distance walked (in feet) as measured by the six minute walk test. Two walk tests were completed at each endpoint visit (separated by 30 min). The average distance of the two walk tests will be used for analysis. The change in this measure over time is assessed using a repeated measures linear regression model of trajectory (change over time). If there is no interaction between change over time and treatment a single calculated value is the slope (the change per six months) from the model. If there is an interaction, the p-value for interaction is presented along with two calculated values representing the slope (the change per six months) for each treatment arm from the model.
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had available analyzable six minute walk test data at baseline, 6 month, and 12 month.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 15
meters | 9.81 (7.53) | -3.43 (5.72)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.583, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase I trial; slope of time = 2.82, Standard Error of Mean 5.06 — "Standard error of the mean" is the standard error of the estimate over time of the slope

24. Secondary Outcome: Change From Baseline in Minnesota Living With Heart Failure Questionnaire Score
Description: Change in the quality of life summary score as measured by the Minnesota Living with Heart Failure Questionnaire. Minimum and maximum scores for scale are 0 and 105 respectively. Lower scores indicative of better outcome.
Time Frame: Baseline to 12 months
Population: Participants who had available analyzable MLHFQ summary score at baseline and 12 month.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 14
score on a scale | -25.45 (25.65) | -12.63 (14.59)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; The change in MLHFQ summary score was compared using ANCOVA analyses adjusting for baseline values; Test type: Superiority; p = 0.048, ANCOVA; Mean Difference (Final Values) = -12.82, 95% CI 2-sided [-30.49 to 4.84], Standard Error of Mean 8.37 — Confidence intervals based on t-test

25. Secondary Outcome: Change From Baseline in Minnesota Living With Heart Failure Questionnaire Score-Trajectory
Description: The change in this measure over time is assessed using a repeated measures linear regression model of trajectory (change over time). If there is no interaction between change over time and treatment a single calculated value is the slope (the change per six months) from the model. If there is an interaction, the p-value for interaction is presented along with two calculated values representing the slope (the change per six months) for each treatment arm from the model.
  Minimum and maximum scores for scale are 0 and 105 respectively. Lower scores indicative of better outcome.
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had available analyzable MLHFQ data at baseline, 6 month, and 12 month.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 14
score on a scale | -10.15 (2.94) | -6.05 (1.92)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0002, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase I trial; slope of time = -8.07, Standard Error of Mean 1.86 — "Standard error of the mean" is the standard error of the estimate over time of the slope

26. Secondary Outcome: Change From Baseline in N-Terminal Pro-Brain Natriuretic Peptide (NT-proBNP)
Description: Change in N-Terminal pro-Brain Natriuretic Peptide (NT-proBNP) as measured via laboratory blood draw
Time Frame: Baseline to 12 months
Population: Participants who had available analyzable NT-proBNP results at baseline and 12 month. Log transformation used. p-values were obtained from transformed data.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 15
pg/ml | -392.58 (953.71) | -76.76 (410.48)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; The change in NT-proBNP was compared using ANCOVA analyses adjusting for baseline values. Data log transformed. p-values were obtained from transformed data; Test type: Superiority; p = 0.199, ANCOVA; Mean Difference (Final Values) = -315.80, 95% CI 2-sided [-947.50 to 315.80], Standard Error of Mean 295 — Confidence intervals based on t-test

27. Secondary Outcome: Change From Baseline in N-Terminal Pro-Brain Natriuretic Peptide (NT-proBNP)-Trajectory
Description: as for outcome 9
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had available analyzable NT-proBNP results at baseline, 6 month, and 12 month. Log transformation used for the regression. p-values were obtained from transformed data.
Measure: Least Squares Mean (Standard Error); unit: pg/ml
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 12 | 15
pg/ml | -184.18 (113.16) | -58.58 (49.41)
Statistical Analysis 1: Comparison: Allo-MSCs vs Placebo; Repeated-measures linear regression models were used to address trajectories (upward or downward trends) over time within each of the treatment groups. If there was no significant interaction, only one trajectory (slope) was reported. Log transformation used for the regression. p-values were obtained from transformed data; Test type: Superiority; p = 0.229, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase I trial; slope of time = -23.391, Standard Error of Mean 202.080 — "Standard error of the mean" is the standard error of the estimate over time of the slope

28. Secondary Outcome: Cumulative Days Alive and Out of Hospital for Heart Failure
Description: Days alive and out of hospital for heart failure during the study evaluation period. Subjects were allotted a visit window extending 30 days past their anticipated 12-month visit (i.e., 395 days).
Time Frame: Baseline to End of 12 Month Visit Window (i.e. 395 days after intervention)
Population: Comparison of the two groups on days alive and out of the hospital for heart failure during the 12 month study evaluation period. Analysis includes all study subjects (including the 6 open label patients).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Allo-MSCs | Placebo
Number analyzed (Participants) | 20 | 16
days | 368 (25.8) | 363 (31.9)

ADVERSE EVENTS:
Time Frame: Events reported are from randomization date to the 12 month endpoint data collection window (i.e 395 days post intervention)
Description: Events were assessed systematically at each study visit during the physical exam assessment. A standard workbook was used to collect event details. Sponsor safety team reviewed events and requested additional documentation as needed.
Arm/Group | Allo-MSCs | Placebo
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/17
Serious Adverse Events (participants affected / at risk) | 5/20 | 11/17
Other Adverse Events (participants affected / at risk) | 4/20 | 4/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allo-MSCs (N=20) | Placebo (N=17)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 2 (3)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular deconditioning (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Chrohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Drug induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Post operative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Lead dislodgement (Product Issues) | 0 (0) | 1 (1)
Device lead damage (Product Issues) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allo-MSCs (N=20) | Placebo (N=17)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 4 (4)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Heterogeneous history of cancer; Lengthy time interval (both from cancer diagnosis and AIC diagnosis); Age of cancer records (>15 yrs in some cases); Natural history of AIC in our cohort better than expected on the basis of the literature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT02509156/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT02509156/Prot_SAP_002.pdf